CLINICAL TRIAL: NCT05002205
Title: Long-term Effects of COVID-19: a Comparative Cohort Study
Acronym: CoCo
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ann Van den Bruel, Associate professor, KU Leuven
Other Study IDs: S65768
Record Dates: First submitted 2021-07-16; First posted 2021-08-12 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19: exposed cohort with a diagnosis of COVID-19 in the last 6 months
  Interventions: Other: Questionnaires; Other: spirometry; Other: ECG; Other: 1 minute sit to stand test; Other: Vital parameters
- no history of COVID-19: non-exposed cohort without a diagnosis of COVID-19. Tested for COVID-19 because of symptoms at the same time (+/- 1 month) as the exposed cohort.
  Interventions: Other: Questionnaires; Other: spirometry; Other: ECG; Other: 1 minute sit to stand test; Other: Vital parameters

INTERVENTIONS:
Other: Questionnaires — Participants will be followed up by means of online surveys and 2 study visits.
Other: spirometry — During two study visits, the lung function will be measured (FVC, FEV1)
Other: ECG — During two study visits, the presence of arrhythmia will be explored.
  Other Names: elecrocardiogram
Other: 1 minute sit to stand test — Physical endurance is tested during 2 study visits.
Other: Vital parameters — blood pressure, pulse, weight

SUMMARY:
This study is a longitudinal cohort study which investigates the effect of COVID-19 in ambulatory care. This study aims to assess the effect of COVID-19 beyond the acute phase, i.e. on long-term symptoms, respiratory and cardiovascular health, use of health services, and quality of life.

DETAILED DESCRIPTION:
This study is a longitudinal cohort study comparing two cohorts. One cohort tested positive for SARS-CoV-2 and the other tested negative for SARS-CoV-2 matched by the timing of testing in the past 6 months. Participants will be observed for two years after their test for COVID-19 with online surveys at different time intervals and face-to-face follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in this study for the exposed cohort with a diagnosis of COVID-19 in the last 6 months must meet all of the following criteria:

1. Aged 18 years or older;
2. Positive result on a rapid Ag test or PCR for SARS-CoV-2 for Covid-19 compatible symptoms a maximum of 6 months before inclusion;
3. Patient is community-dwelling;
4. Participant or their proxy is willing and able to give informed consent for participation in this study;
5. Participant is willing to comply with all study procedures.

Participants are sampled in the same practices as the exposed cohort and are eligible for inclusion in this study for the non-exposed without a diagnosis of COVID-19 in the last 6 months when they meet all of the following criteria:

1. Aged 18 years or older;
2. Tested because of suggestive symptoms with a rapid Ag test or PCR for SARS-CoV-2 at the same time (+/- 1 month) as the exposed cohort, of which the result was negative
3. Patient is community-dwelling;
4. Participant or their proxy is willing and able to give informed consent for participation in this study;
5. Participant is willing to comply with all study procedures.

Exclusion Criteria:

Participants eligible for the cohort with COVID-19 in the last 6 months must not meet any of the following criteria:

1. Patients in palliative care;
2. Patients for whom there is already someone from the same household participating;
3. Judgement of the recruiting clinician deems participant ineligible.

Participants eligible for the cohort without COVID-19 must not meet any of the following criteria:

1. A positive test for a SARS-CoV-2 infection in the last 2 years;
2. Patients in palliative care;
3. Patients for whom there is already someone from the same household participating;
4. Judgement of the recruiting clinician deems participant ineligible.

Prior vaccination against Covid-19 is not an exclusion criterion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2 cohorts of people who experienced an infection in the past 6 months of which 1 group had a proven covid-19 infection and 1 group definitely did not.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-08-31 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue severity 6 months after diagnosis of COVID-19. | 6 months post-COVID
  Data for this endpoint are collected with a questionnaire during the first study visit at 6 months. The severity of fatigue will be assessed using the Fatigue Severity Scale (FSS). This is a 9-item scale which measures the severity of fatigue and how it affects a person's activities and lifestyle.
  The score ranges from 7 to 63, with higher values indicating more fatigue.

SECONDARY OUTCOMES:
Incidence of post-COVID symptoms | 6 months, 9 months, 1 year, 1.5 year and 2 years post-COVID
  Incidence of each individual symptoms at 6 months, 9 months, 1 year, 1.5 years and 2 years including cough, difficulty breathing, tightness on the chest, pain in the lungs, throatache, muscle ache, muscle weakness, joint pain, pain between the shoulder blades, headache, dizziness, confusion, concentration loss/lack of focus, concentration problems on short and long term, feeling absent, difficulties finding words/afasia, palpitations, hot flushes, sleeping problems, abdominal pain, blurred vision, nerve pains, sensory disorders, mood swings, anxiety, depressive feeling (Source: questionnaire during study visits and remote surveys)
Participants' quality of life | 6 months, 9 months, 1 year, 1.5 year and 2 years post-COVID
  Euroqol EQ-5D-5L: The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems, where higher scores indicate a better outcome (Source: questionnaire during study visits and remote surveys)
Lung function (FEV1, FVC) | 6 months and 1 year post-COVID
  (Source: spirometry during study visits at 6 months and 1 year)
The degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4 (mMRC scale) | 6 months, 9 months, 1 year, 1.5 year and 2 years post-COVID
  0, no breathlessness except on strenuous exercise; 1, shortness of breath when hurrying on the level or walking up a slight hill; 2, walks slower than people of same age on the level because of breathlessness or has to stop to catch breath when walking at their own pace on the level; 3, stops for breath after walking ∼100 m or after few minutes on the level; and 4, too breathless to leave the house, or breathless when dressing or undressing
Gustatation | 6 months, 9 months, 1 year, 1.5 year and 2 years post-COVID
  scale from 1 to 10; higher scores indicate more problems with gustation. (Source: questionnaires during study visits and remote surveys)
Olfaction | 6 months, 9 months, 1 year, 1.5 year and 2 years post-COVID
  scale from 1 to 10; higher scores indicate more problems with olfaction. (Source: questionnaires during study visits and remote surveys)
Incidence of diagnoses of COPD | 6 months and 1 year post-COVID
  Source: spirometry during study visits
Exercice capacity and endurance | 6 months and 1 year post-COVID
  Source: 1 minute sit to stand test during study visits
Incidence of cardiovascular events including AMI, lung embolism of stroke | 6 months and 1 year post-COVID
  Questionnaire during study visits
Number of Unplanned hospital admissions of at least 24 hours | within 2 years post-COVID
  Source: questionnaire during study visits and remote surveys
Number of Visits to healthcare professionals | within 2 years post-COVID
  Source: questionnaire during study visits and remote surveys
Number of days absent from work | within 2 years post-COVID
  Source: questionnaire during study visits and remote surveys
Exploring treatments attempted by patients in the scope of post-COVID symptoms | within 2 years post-COVID
  Categorical options: no treatment; vitamines; antibiotics; puffs; pain medication; anti-inflammatory drugs; others Source: questionnaire during study visits and remote surveys
Exploring the type of counseling patients with post-covid symptoms use. | within 2 years post-COVID
  Categorical options: no counseling; psychologist; physiotherapist; GP; rehabilitation doctor; other Source: questionnaire during study visits and remote surveys
Exploring the meaning of fatigue post-COVID and its impact on their daily lives | +/- 6 months post-COVID
  Source: semi-structured interviews online

IPD SHARING:
Plan to Share IPD: Undecided